CLINICAL TRIAL: NCT04022356
Title: Validity of Using Connected Soles In Measuring Steps Number In the Older Subject, Hospitalized in Follow-up and Rehabilitative Care and Achieve Its Rehabilitation Objectives
Acronym: SEMCOPAGE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was not able to start within the time limit due to Coronavirus
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018-A03468-47
Record Dates: First submitted 2019-05-09; First posted 2019-07-17 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Patient Recovering Maximum Walking Capacity, Over 10 Meters
Keywords: counting; steps; Connected Soles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connected soles (Experimental): Number of steps recorded by the soles (activation per smartphone)
  Interventions: Device: Feetme Connected Soles
- Gold Standard (Active Comparator): Number of steps counted by two observers viewing the film
  Interventions: Device: Feetme Connected Soles

INTERVENTIONS:
Device: Feetme Connected Soles — Walk for 10 meters (and 30meters):
  * By wearing the European Community (EC) labelled connected soles in patient's shoes, triggered by smartphone- collection of data by smartphone
  * By being filmed by a camera camera mounted on a tripod (excluding the face) for steps counting (2 observers).
  If there is a technical problem during the walk test, this one can be performed 1 time again 1 hour after initial test.This is expected to happen very rarely.

SUMMARY:
The purpose of this study is to evaluate counting steps by connected soles worn in the shoes of subjects, having recovered the maximum walking capacities of patients . To answer the question asked in the study, it is planned to include 60 patients over 70 years of age.

DETAILED DESCRIPTION:
The main objective of this interventional, monocentric, transverse, nonrandomized and prospective study is to assess the concordance of step counting between connected soles and video, in elderly subjects hospitalized in Follow-up and rehabilitation care, at Paul Brousse hospital, having recovered maximum walking capacities of participants, on 10 meters.

After inclusion, following data will be collected : Measure blood pressure, heart rate, neurological and cardiological exam, pneumological exam, Short Physical Performance Battery Score

Feetme connected soles comply with European standards (CE label no. 29762). The study will consist of 10-metre walk for patient during a rehabilitation session :

* By wearing the soles connected to patient's size (in patient's usual shoes). The recording of data will be triggered by an investigator, via an application downloaded on a smartphone. The application will trigger and stop the registration of soles.
* While being filmed by a camcorder mounted on a tripod (excluding the face) for footsteps.

The test will be filmed (excluding the face) to avoid a measurement bias in counting steps. Two physician observers will view each patient's film in a second time in order to perform the step count.

Before starting the walk, an on-site observer will ensure that the footings are set to 0 for counting step and that the recording is stopped after 10 metres.

If this is deemed possible by the referring physiotherapist, the same protocol will then be carried out over 30 meters (new test: the patient who can do it will perform 40 meters in total (10 meters then test of 30 meters).

ELIGIBILITY:
Inclusion Criteria:

* Age >70 years olde
* Patients able to walk 10 meters
* Patients who received physiotherapy
* Patients able to understand instructions and freely consent (mini mental state examination (MMSE) ≥ 20
* Informed consent, major unprotected
* Membership in a social security scheme

Exclusion Criteria:

* Unable to walk the required distance (severe dyspnea, post-fall syndrome, blindness)
* Foot sores (bedsores or other)
* Patients participating in another intervention study
* Major patients protected or deprived of study freedom

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of steps number to cover the distance of 10 meters according connected soles | 3 days
  The main evaluation criterion is the number of steps taken by the patient to travel the distance of 10 meters. A ground marking will be done using a tape meter to highlight the distance of 10 meters.The number of steps will be counted using the connected soles and video. The soles count the step thanks to the foot pressure and the data are collected on smartphone. A video will be recorded simultaneously (fluted face) during the walk.

SECONDARY OUTCOMES:
Assessment of steps number to cover the distance of 30 meters according connected soles and video | 3 days
Assessment of soles comfort according Likert scale | 3 days

IPD SHARING:
Plan to Share IPD: Undecided